CLINICAL TRIAL: NCT02275897
Title: Injection Speed of Spinal Anaesthesia for Asian Women Undergoing Lower Segmental Caesarean Section and the Incidence of Hypotension and/or Use of Vasopressors
Brief Title: Effect of Different Injection Speeds for Spinal Anaesthesia in Caesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ministry of Health, Malaysia (Other Government)
Responsible Party: Principal Investigator, Dr. Chiang CF, Medical Officer, Ministry of Health, Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NMRR-13-608-16854 (IIR)
Record Dates: First submitted 2014-10-15; First posted 2014-10-27 (Estimated); Last update posted 2014-12-12 (Estimated); Status verified 2014-12

CONDITIONS: Pregnancy; Effects of; Anesthesia, Spinal and Epidural; in Pregnancy
Keywords: Lower Segmental Caesarean Section (LSCS); Speed of Injection; Spinal Anaesthesia; Anesthesia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Slow Speed (Experimental): Slow group patients will receive spinal injection over 60 seconds. Vital signs monitored every minute after injection. Hypotension is treated with IV Phenylephrine or Ephedrine.
  Interventions: Procedure: Slow Speed of spinal injection
- Fast Speed (Experimental): Fast group patients will receive spinal injection over 15 seconds. Vital signs monitored every minute after injection. Hypotension is treated with IV Phenylephrine or Ephedrine.
  Interventions: Procedure: Fast Speed of spinal injection

INTERVENTIONS:
Procedure: Slow Speed of spinal injection — Speed of injection over 60 seconds
  Arms: Slow Speed
Procedure: Fast Speed of spinal injection — Speed of injection over 15 seconds
  Arms: Fast Speed

SUMMARY:
The purpose of this study is to investigate if prolonging the speed of injection during spinal anaesthesia can reduce the incidence of hypotension and/or medication requirements thereby making it safer for the mother and foetus.

DETAILED DESCRIPTION:
We plan to investigate if by varying the speed of injection during spinal anaesthesia, will there be a difference in the incidence of hypotension. Hypotension is a common complication especially for pregnant women undergoing caesarean section. A high speed of injection can theoretically cause a higher spread of anaesthetic, which may increase the incidence of hypotension. We want to know if by prolonging the injection time, will this lead to a reduction in a rate of hypotension.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* singleton term pregnancy
* American Society of Anesthesiologists (ASA) class I-II

Exclusion Criteria:

* Severe pre-eclampsia
* contraindications to spinal anaesthesia
* Height <150cm or >180cm
* Weight ≥100kg
* Baseline systolic BP <90 mmHg
* Baseline systolic BP >150mmHg
* Category 1 urgency for delivery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2013-03; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Incidence of Hypotension | First 10 minutes after injection
  How many patients will experience a drop in systolic Blood Pressure of greater than 20%

SECONDARY OUTCOMES:
Use of vasoconstrictors | First 10 minutes after injection
Adequacy of block | Time of surgery
  To determine if the anaesthetic is adequate for the surgery (no pain or movement experienced around the surgical field)

CONTACTS AND LOCATIONS:
Overall Officials: Chun Fai Chiang, MBBS, Principal Investigator — Ministry of Health, Malaysia
Locations (1):
- Hospital Tengku Ampuan Rahimah, Klang, Selangor, Malaysia

REFERENCES:
- [Derived] Chiang CF, Hasan MS, Tham SW, Sundaraj S, Faris A, Ganason N. Injection speed of spinal anaesthesia for Caesarean delivery in Asian women and the incidence of hypotension: A randomised controlled trial. J Clin Anesth. 2017 Jun;39:82-86. doi: 10.1016/j.jclinane.2017.03.025. Epub 2017 Apr 1. PMID 28494915